CLINICAL TRIAL: NCT06926283
Title: A Phase I, Open-Label, Multicenter, First-in-Human, Dose Escalation and Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profiles and Preliminary Efficacy of DXC008 in Patients With Prostate Cancer and Other Solid Tumors (Such as Ewing Sarcoma)
Brief Title: A Study of DXC008 in Patients With Prostate Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou DAC Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DXC008-001
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Other Solid Tumors; Ewing Sarcoma
MeSH Terms: conditions — Prostatic Neoplasms; Sarcoma, Ewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DXC008 (Experimental)
  Interventions: Drug: DXC008

INTERVENTIONS:
Drug: DXC008 — Cohort A: Once every 2 weeks (Q2W) with a cycle length of 14 days. Cohort B: Once every 3 weeks (Q3W) with a cycle length of 21 days.

SUMMARY:
This is a phase I, open-label, first-in-human clinical study designed to evaluate the safety, tolerability, MTD, DLT, RP2D, the PK characteristics, preliminary anti-tumor activity, the immunogenicity of DXC008 in patients with prostate cancer and other solid tumors such as Ewing sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily sign the ICF and follow the protocol requirements.
2. Male or female.
3. Age: ≥ 18 years and ≤ 75 years.
4. Expected life expectancy ≥ 6 months.
5. ECOG performance status score: 0-2.
6. Patients with various solid tumors who have failed standard treatment, including but not limited to progressive mCRPC.
7. Serum testosterone level during screening and prior to the first dose of investigational product: ≤50 ng/dL (≤1.73 nmol/L).
8. Cohort 1: at least one measurable lesion as defined by RECIST v1.1. Cohort 2: at least one metastatic lesion on CT/MRI, or bone scan imaging at baseline. Patients are assigned to the appropriate cohort as assessed by the investigator, the study procedures in Cohort 1 and Cohort 2 may be performed in parallel and simultaneously, it is not necessary to wait until all procedures in either cohort have been completed before initiating procedures in the other cohort.
9. Toxicities from prior antitumor therapy must have recovered to Grade ≤ 1 as defined in the NCI-CTCAE v5.0 (except alopecia), or Grade 2 as defined by NCI-CTCAE v5.0, except for toxicity not constituting a safety risk by investigator judgment (eg, Grade 2 peripheral neurotoxicity).
10. Organ function of the subjects must meet the following requirements:

Hematology:

1. ANC ≥ 1.5 × 10^9/L (prior use of G-CSF is allowed, but G-CSF use is not allowed within 7 days prior to the screening laboratory tests).
2. Platelet count ≥100×10^9/L (platelet transfusion is not allowed within 7 days before the screening laboratory tests).
3. HGB ≥ 90 g/L (RBC transfusion or recombinant human erythropoietin use is allowed; RBC transfusion is not allowed within 7 days prior to the screening laboratory tests).

Liver function:

1. Total bilirubin (TBIL) ≤1.5×ULN, except for subjects with congenital bilirubinemia, such as Gilbert syndrome (direct bilirubin ≤1.5×ULN).
2. AST and ALT ≤ 3.0 × ULN. For patients with liver metastases, both AST and ALT ≤5×ULN.

Renal function:

Ccr ≥ 60 mL/min; or creatinine ≤ 1.5 × ULN; urinalysis results show protein urine ≤ 1 +.

For subjects with urine protein ≥2+ in urinalysis during the screening period, a 24-hour urine protein quantification should be performed, and those with 24-hour urine protein quantification ≤1 g can be enrolled.

Coagulation function:

1. INR≤1.5.
2. APTT or PT ≤ 1.5 × ULN. LVEF≥50%. 11.Subjects and their spouses agree to use effective instrumental or pharmacologic contraception (excluding safe period contraception) from the time of ICF signing until 6 months after the last dose of investigational product.

Exclusion Criteria:

1. Within 14 days prior to the first dose: Have undergone plasmapheresis, treated with prednisone at > 10 mg/day for > 3 consecutive days or equivalent dose of systemic corticosteroids or equivalent anti-inflammatory medication (Those who have received short-term treatment with such medications for the prevention of contrast media allergy may be enrolled).
2. Have received systemic antineoplastic therapy or investigational product treatment within 28 days or 5 half-lives (whichever is shorter) prior to the first dose, have received radiotherapy within 14 days prior to the first dose.
3. Have received monoclonal antibody treatment within 30 days prior to the first dose.
4. History of solid organ transplantation.
5. Prior treatment with XXX-targeted therapy or topoisomerase inhibitors (in Phase Ia clinical study only).
6. Presence of meningeal or brain metastases.
7. Evidence of cardiovascular risk, including any of the following:

   1. QTcF interval ≥ 470 msec (QT interval must be corrected for heart rate using the Fridericia formula [QTcF]).
   2. Evidence of current clinically significant untreated arrhythmias, including clinically significant ECG abnormalities including second-degree (Mobitz Type II) or third-degree atrioventricular (AV) block.
   3. Within 6 months before screening, history of myocardial infarct, acute coronary syndrome (including unstable angina pectoris), coronary angioplasty or stent implantation, or bypass grafting.
   4. Class III or IV heart failure - as defined by the New York Heart Association Functional Classification.
   5. Uncontrolled severe hypertension: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥ 100 mmHg.
8. Have dyspnea or any current condition that needs continuous oxygen therapy, or current active pneumonia or interstitial lung diseases (except mild cases as judged by the investigator).
9. History of other primary malignancies, except for the following: malignancies that have been cured and have a very low risk of recurrence within 5 years, such as basal cell carcinoma and squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast.
10. Have severe unhealed wound, ulceration or bone fracture, or have received major surgery within 28 days prior to administration or expected major surgery during the clinical study.
11. Prior history of allergy to any component or excipient of DXC008.
12. Active hepatitis B with HBV-DNA greater than central upper limit of normal or greater than 1000 copies/mL, active hepatitis C (Hepatitis C virus antibody positive with HCV RNA greater than lower limit of detection value).
13. Known to be seropositive for the HIV; have active syphilis (only patients with a positive syphilis antibody are eligible for enrollment in the study), possible presence of active tuberculosis (chest imaging within 3 months prior to the first dose indicates active tuberculosis infection).
14. Patients with active bleeding within 30 days before screening, or, judged by the investigator, to be at risk of massive digestive tract hemorrhage, hemoptysis, etc.; or with hereditary bleeding tendency or coagulation disorder, or bleeding symptoms requiring other medical intervention.
15. Have experienced serious arterial/venous thrombosis events within 6 months prior to the first dose, such as cerebrovascular accident (including transient cerebral ischemic attack), deep venous thrombosis, pulmonary embolism.
16. Female subjects with positive serum pregnancy test or who are breastfeeding.
17. Those with active infection requiring drug intervention (CTCAE ≥ Grade 2) within 2 weeks prior to the first dose of study treatment, uncontrollable pleural effusion, ascites, pericardial effusion requiring repeated drainage.
18. Have received vaccination with live attenuated vaccine within 28 days prior to the first dose or planned to receive such vaccination during the study period.
19. Patients with other conditions judged by the investigator that may have adverse effect on the patient's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants that experienced dose limiting toxicities(DLTs) at given dose level. | 28 days
  Dose Limiting Toxicities (DLTs) In Order to Determine the Maximum Tolerated.
Number of participants with adverse events (AEs). | After first infusion of study drug, Through study completion an average of 1 year.
  The adverse events will be evaluated in accordance with CTCAE v5.0. The investigator shall assess the relationship between the events and investigational product.

SECONDARY OUTCOMES:
Maximum observed serum or plasma concentration (Cmax). | Through study completion an average of 1 year.
  One of the pharmacokinetics parameters for DXC008 investigator shall assess the relationship between the events and investigational product.
Maximum serum drug time (Tmax). | Through study completion an average of 1 year.
  One of the pharmacokinetics parameters for DXC008.
Apparent volume of distribution(Vd). | Through study completion an average of 1 year.
  One of the pharmacokinetics parameters for DXC008.
Measurement of objective response rate (ORR) per RECIST 1.1. | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
  Percentage of subjects achieving complete response (CR) or partial response (PR).
ORR per Prostate Cancer Working Group 3 (PCWG3). | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year.
  Percentage of subjects achieving complete response (CR) or partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Zhisong He, Principal Investigator — Peking University First Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No